CLINICAL TRIAL: NCT05721313
Title: Vital Root Amputation in Molars With Advanced Periodontal Furcation Involvement: a Preliminary Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azienda Ospedaliera, Universitaria Policlinico Vittorio Emanuele (Other)
Responsible Party: Principal Investigator, Giovanni Barbagallo, DDS, DMD, Azienda Ospedaliera, Universitaria Policlinico Vittorio Emanuele
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COM
Record Dates: First submitted 2023-01-25; First posted 2023-02-10 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Periodontal Diseases; Furcation Defects
Keywords: Periodontal disease; Furcation defects; Root resection
MeSH Terms: conditions — Periodontal Diseases; Furcation Defects | interventions — Apicoectomy

STUDY DESIGN:
Intervention Model Description: Pilot cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with advanced periodontal furcation involvement (Experimental)
  Interventions: Procedure: root resection

INTERVENTIONS:
Procedure: root resection — It will be carried out under local anestesia. Intra-crevicular or para-marginal gingival incision will be carried out and full-tickness mucoperiostal flaps will be raised to expose the affected roots. Whit the use (if possible) of a surgical stent an incision will be performed on the root to be removed. Biodentine will be used for retrogade obturation. The flaps will be sutured.

SUMMARY:
The goal of this clinical trial is to test in 10 patients with advanced furcation involvement on molars. The main question[s] it aims to answer are:

• Is it possible to carry out root resection without endodontic treatment on molars? Tooth vitality will be checked (positive response to cold test). Root resection will be carried out under local anestesia.

Following visits will be carried out for re-evaluation/maintenance according to clinical care every 3 mounths until 3 years follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with stage III-IV periodontitis
* Compliantpatient, as shown by full mouth plaque score<30%
* Previous non-surgical periodontal therapy within 6 mounths
* Maxillary or mandibular molar affected by periodontal furcation involvement and scheduled for root resection
* Positive to sensibility testing (cold/electric pulp tests)
* No prosthesis or large restorations
* Sufficiently divergent roots to make root resection feasible
* Root trunk lenght at 3 mm as measured in periapical radiograph

Exclusion Criteria:

* Systemic contraindications to perform periodontal surgery/root resection
* Fused roots
* Presence of periapical radiolucency
* Furcation class III affecting all roots of maxillary molar

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
Tooth vitality (positive response to cold test) | 3-year follow-up
  following the 3rd visit will be make a re-evaluation of the tooth vitality, by a positive response to cold test, every 3 month.
No periapical lesion | 3-year follow-up
  following the 3rd visit will be make a re-evaluation of the periapical heath condition, by a periapical rx, every year

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Odontoiatrico Mediterraneo, Catania, CT, Italy